CLINICAL TRIAL: NCT02747758
Title: Randomized Controlled Clinical Trial Evaluating Transcranial Direct Current Stimulation (tDCS) in Chronic Pain Patients With Neuropathy
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Chronic Neuropathy
Acronym: Neuro-tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment due to CORONA
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Tafelski, physician scientist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neuro-tDCS1
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Neuropathic Pain; Neuralgia
Keywords: neuropathic pain; neuralgia; tDCS; transcranial direct current stimulation
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Sham Comparator): sham transcranial direct current stimulation (tDCS)
  Interventions: Device: sham transcranial direct current stimulation (tDCS)
- cathodal stimulation (Experimental): cathodal transcranial direct current stimulation (tDCS)
  Interventions: Device: cathodal transcranial direct current stimulation (tDCS)
- anodal stimulation (Experimental): anodal transcranial direct current stimulation (tDCS)
  Interventions: Device: anodal transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: cathodal transcranial direct current stimulation (tDCS) — transcranial direct current stimulation (tDCS) is applied in active groups using cathodal active M1 stimulation. Active stimulation is applied with 2mA direct current via 20cm² electrodes.
  Arms: cathodal stimulation
Device: sham transcranial direct current stimulation (tDCS) — transcranial direct current stimulation (tDCS) is applied in active groups using a sham-stimulation including ramp up and ramp down of current.
  Arms: Control
Device: anodal transcranial direct current stimulation (tDCS) — transcranial direct current stimulation (tDCS) is applied in active groups using anodal active M1 stimulation. Active stimulation is applied with 2mA direct current via 20cm² electrodes.
  Arms: anodal stimulation

SUMMARY:
This study evaluates the effect of additional transcranial direct stimulation (tDCS) on pain in patients with chronic neuropathic pain undergoing treatment with regional anaesthesiological techniques.

DETAILED DESCRIPTION:
About 3.8 Million persons in Germany suffer from chronic pain with a relevant physical and social impairment representing approximately 7% of the population. Chronic pain conditions include patients with neuropathic pain such as trigeminal neuralgia, post-zoster pain or pain after amputations. There is a significant number of patients with pain without response to optimised drug therapy. Especially in these chronic pain patients there is data demonstrating maladaptive plasticity as pathophysiological evidence of structural changes in brain connectivity. Patients are treated with multimodal pain therapy concepts including interventional procedures with nerve infiltration techniques.

One innovative therapeutic option for pain patients is transcranial direct current stimulation (tDCS): In recent clinical trials, patients reported on reduced overall pain intensity following tDCS stimulation series shown e.g. from Bolognini et al., Antal et al. and most recently from Volz and colleagues. However, there is no current data available evaluating a role of tDCS for patients with chronic neuropathic pain treated with regional anaesthesiological techniques.

Objective: To evaluate effect of additional tDCS series on pain in patients with chronic neuropathic pain

Primary study endpoint: relative reduction in pain (initial VAS measured versus VAS after completion of the therapy series) as a numeric value between 0 and 10.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuropathic pain with indication of regional anaesthesiological interventions

Exclusion Criteria:

* <18 years of age
* Pregnancy
* Police custody
* Epilepsy
* Participation in another prospective clinical intervention study within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
relative pain intensity | after completion of therapy series, typically after 2 weeks of treatment
  relative reduction in pain intensity (initial VAS measured versus VAS after completion of the therapy series), VAS as a numeric value between 0 and 10.

SECONDARY OUTCOMES:
acute pain reduction by tDCS application (relative reduciton measured as VAS after completion of tDCS stimulation versus initial VAS measured before stimulation) | 30 Minutes after application
  relative reduction of pain intensity before and after each tDCS session and infiltration
time to next regional-anesthesiological series | 6 months
  time until patients need additional regional-anesthesiological interventions
number of regional-anesthesiological interventions for pain control | 10 days
  number of required regional-anesthesiological interventions to achieve sufficient pain reduction
adverse events | 1 months
  Analysis of adverse reaction (skin redness, headache, concentration, other)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schäfer, Prof. MD, Study Chair — Charité University Berlin
Locations (1):
- Pain Clinic of Charité hospital Campus Virchow Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tafelski S, Beutlhauser T, Gouliou-Mayerhauser E, Fritzsche T, Denke C, Schafer M. [Practice of regional anesthesia for chronic pain patients in specialized pain services : A nationwide survey in Germany]. Schmerz. 2015 Apr;29(2):186-94. doi: 10.1007/s00482-014-1503-6. German. PMID 25479710
- [Background] Flor H, Nikolajsen L, Staehelin Jensen T. Phantom limb pain: a case of maladaptive CNS plasticity? Nat Rev Neurosci. 2006 Nov;7(11):873-81. doi: 10.1038/nrn1991. PMID 17053811
- [Background] Hauser W, Schmutzer G, Hinz A, Hilbert A, Brahler E. [Prevalence of chronic pain in Germany. A representative survey of the general population]. Schmerz. 2013 Feb;27(1):46-55. doi: 10.1007/s00482-012-1280-z. German. PMID 23321703
- [Background] Antal A, Terney D, Kuhnl S, Paulus W. Anodal transcranial direct current stimulation of the motor cortex ameliorates chronic pain and reduces short intracortical inhibition. J Pain Symptom Manage. 2010 May;39(5):890-903. doi: 10.1016/j.jpainsymman.2009.09.023. PMID 20471549
- [Background] Volz MS, Farmer A, Siegmund B. Reduction of chronic abdominal pain in patients with inflammatory bowel disease through transcranial direct current stimulation: a randomized controlled trial. Pain. 2016 Feb;157(2):429-437. doi: 10.1097/j.pain.0000000000000386. PMID 26469395
- See also: Pain Clinic Website — https://anaesthesieintensivmedizin.charite.de/leistungen/schmerztherapie/
- Available data/document: Clinical Study Report — https://www.frontiersin.org/articles/10.3389/fneur.2023.1069434/full — The research report is published open access: ORIGINAL RESEARCH article Front. Neurol., 01 March 2023, Volume 14 - 2023 | https://doi.org/10.3389/fneur.2023.1069434